CLINICAL TRIAL: NCT03551756
Title: Assessment of Biomarkers in Patients With Decompensated Heart Failure and Underlying Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CirQuest Labs, LLC (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CQ 17-11-009
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure & Coronary Artery Disease: Biomarker assessment in adults with decompensated heart failure and significant underlying coronary artery disease
  Interventions: Other: Biomarker Assessment
- Healthy Adult: Biomarker assessment in 20 healthy age-matched subjects
  Interventions: Other: Biomarker Assessment

INTERVENTIONS:
Other: Biomarker Assessment — Exploratory Biomarker Analysis for cardiac patients versus healthy adults

SUMMARY:
Assessment of Biomarkers in Patients with Decompensated Heart Failure and Underlying Coronary Artery Disease

DETAILED DESCRIPTION:
This is a cross-sectional, single center exploratory study of plasma biomarker levels in adults with decompensated heart failure and significant underlying coronary artery disease as compared with age-matched healthy controls. Subjects will not receive a therapeutic treatment as part of this study and will undergo a single blood draw.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Heart Failure with Coronary Artery Disease Subjects

* Symptomatic heart failure (≥ 3 months) with most recently documented LVEF ≤ 40% (Echo must have been completed in last 12 months prior to enrollment.)
* Significant underlying coronary artery disease as evidenced by:
* previous myocardial infarction
* prior coronary artery bypass graft
* 50% coronary stenosis of one or more arteries and/or
* history of percutaneous coronary intervention with or without stenting
* Age 18 years or older at the first screening visit

Group 2: Healthy Subjects

• Age 18 years or older at the first screening visit and within 20% of mean age of Group 1 Subjects

Exclusion Criteria:

Group 1:

* Documented history of "severe" valvular disease
* Documented history of atrial fibrillation, ventricular fibrillation or ventricular tachycardia.
* Recent or current use of anticoagulant medications such as fXa inhibitors, direct thrombin inhibitors, vitamin K antagonists, or heparin. (within 1 month of screening)

Group 2:

* Known significant cardiovascular or hematological condition
* Recent or current use of anticoagulant medications such as fXa inhibitors, direct thrombin inhibitors, vitamin K antagonists, or heparin. (within 1 month of screening)
* Recent cold or flu symptoms, respiratory infection or surgery (within 2 weeks of screening)
* History of Asthma
* History of peptic ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects with the study diagnosis and 20 healthy age-matched subjects, no restrictions on gender, race, or ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Biomarker assessment | 1 day
  Exploratory biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K. Jennings, PhD, Principal Investigator — CirQuest Labs, LLC
Locations (3):
- United States (3):
  - University of Florida, Jacksonville, Florida
  - Stern Cardiovascular, Germantown, Tennessee
  - CirQuest Labs, LLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided